CLINICAL TRIAL: NCT00180076
Title: Efficacy and Safety of Budesonide in Maintenance Treatment of Collagenous Colitis
Brief Title: Budesonide for Maintenance Treatment of Collagenous Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIMIC
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Collagenous Colitis
Keywords: collagenous colitis; microscopic colitis; budesonide
MeSH Terms: conditions — Colitis, Collagenous; Colitis, Microscopic | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
The purpose of this study is to determine whether orale budesonide is effective in maintaining clinical remission in patients with collagenous colitis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether orale budesonide is effective in maintaining clinical remission in patients with collagenous colitis.

ELIGIBILITY:
Inclusion Criteria:

* collagenous colitis
* diarrhea
* written informed consent

Exclusion Criteria:

* infectious causes for diarrhea
* other inflammatory bowel diseases
* history of colonic surgery
* celiac disease
* malignancies
* severe concomitant diseases
* use of budesonide, steroids, mesalazine within the previous 2 weeks
* known intolerance to budesonide
* history of lack of response to budesonide
* pregnancy,lactation
* drug and/or alcohol abuse
* lack of compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2008-03

PRIMARY OUTCOMES:
Proportion of patients in clinical remission after 6 months

SECONDARY OUTCOMES:
time to relapse
safety
quality of life
histological improvement

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, Prof., Principal Investigator — Medical Department I, Technical University Hospital, Dresden, Germany
Locations (1):
- Medical Department I, Technical University Hospital, Dresden, Germany